CLINICAL TRIAL: NCT04734145
Title: Breathprinting (e-Nose) Technology for the Identification of Early-Stage Lung Cancer
Brief Title: Using e-Nose Technology to Identify Early Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-349
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Lung; Node; Lung Cancer
Keywords: lung cancer; lung nodule; lung node; Memorial Sloan Kettering Caner Center; 20-349; Breathprinting
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with an Undiagnosed Pulmonary Nodule: One hundred evaluable individuals aged 21 to 85 years with a single undiagnosed pulmonary nodule measuring <3 cm, clinically staged as cT1N0M0 (eighth edition of the TNM staging manual) by CT and PET scans, will be enrolled in this diagnostic study and will undergo e-nose testing. These patients must have a risk assessment profile that, according to institutional guidelines, identifies them as candidates for subsequent surgical resection of the pulmonary nodule, which will confirm the results of the breathprinting analysis.
  Interventions: Diagnostic Test: Breathprinting test

INTERVENTIONS:
Diagnostic Test: Breathprinting test — Consented, enrolled participants will undergo a breathprinting test (e-nose) during the presurgical visit and at the same facility as their presurgical or prebiopsy visit, before any attempt is made to obtain cytohistological diagnosis of the pulmonary nodule.
  Other Names: E-Nose

SUMMARY:
The purpose of this study is to test the ability of a new technology called breathprinting, or electronic nose (e-nose), to detect early-stage lung cancer. Additionally, researchers also want to see if the e-nose technology is more effective at diagnosing lung cancer if the tumor size is larger.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-85
* Single, monolateral nodule of at least 50% solid composition visible on chest CT scan (with or without contrast) suspicious for lung cancer.
* MSK radiologist report or read suggestive (i.e. at least 50% certainty) of suspected primary lung cancer (in accordance with the level of certainty criteria set forth by MSKCC Radiology)

  o Patients with biopsy-proven early stage, primary lung cancer that meets staging requirements, do not need to also have a radiology report meeting inclusion criteria
* Negative test for COVID-19 performed locally or at MSK, done as part of standard of care testing (i.e. only when required by specific institutional policy) prior to biopsy or surgical procedure
* Eligible for fine-needle aspiration biopsy, robotic bronchoscopy, and/or surgical resection for diagnosis (i.e., does not have comorbidities precluding these).
* Documented, signed, and dated informed consent, obtained before any procedures, for the proposed research study

  o Patient must agree to undergo fine-needle aspiration biopsy, robotic bronchoscopy, and/or surgical resection for diagnosis prior to e-nose collectionNote: Biopsy-proven patients that meet eligible staging criteria who are not further surgical candidates will be collected prior to next step in standard of care treatment
* Patients with biopsy-proven clinical stage I lung cancer are eligible if the biopsy is done within 6 weeks of the consent date

Exclusion Criteria:

* Age <21 and >85 years at first outpatient visit.
* Multiple ipsilateral or bilateral nodules reported on chest CT scan and/or concurrent as suspicious for lung cancer (note: nodules deemed indeterminate, inflammatory, etc. will not exclude a patient from participating in this study) semisolid GGOs.
* Lung nodule of interest is less than 50% solid in composition
* Per MSK radiologist report or read, the lung nodule of interest is "less likely" or "unlikely" (i.e. less than 50% certainty) to be neoplastic (in accordance with the level of certainty criteria set forth by MSKCC Radiology)
* Any previous history of lung cancer
* History of any non-lung cancer(s) that is currently being treated (note: prior history of completely treated non-lung cancer from any time will be eligible)
* Metastatic lung cancer disease seen on chest CT or PET scan at hilar/mediastinal nodes or contralateral lung or extrathoracic sites.
* Previous medical history of a lung biopsy/surgical procedure for cancer diagnosis (note: patients who underwent a lung biopsy over three years ago that showed negative for lung cancer and patients who underwent a lung biopsy confirming stage I lung cancer within the past 6 weeks will be eligible)

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the principal investigator (PI), or the research team at MSK. If the PI is a member of the treatment team, he or she will screen his or her patients' medical records for suitable research study participants, and discuss the study and the patient's potential for enrolling in the research study with the patient. Potential subjects contacted by their treating physician will be referred to the PI/research staff to record appropriate contact information, so that these patients can be approached about enrolling in the study.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Disease status determined by e-nose testing | up to 1 month (time to biopsy)
  For each study participant, disease status will be determined by e-nose testing ("cancer" or "no cancer") and by TTNA or surgery ("true" status).

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Rocco, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only ), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Study Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org